CLINICAL TRIAL: NCT06120400
Title: Cardiovascular Effects of a Healthy Dietary Pattern Containing Eggs: a Controlled-feeding Study
Brief Title: Cardiovascular Effects of a Healthy Dietary Pattern Containing Eggs
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Penn State University (Other)
Collaborators: American Egg Board (Other)
Responsible Party: Principal Investigator, Kristina Petersen PhD, APD, FAHA, Associate Professor, Penn State University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: HDE
Record Dates: First submitted 2023-11-02; First posted 2023-11-07 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: Cardiovascular Diseases
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Healthy Diet + Eggs (HD+E) (Experimental): 2020-2025 Dietary Guidelines for Americans adherent dietary pattern containing 2 eggs/day/2000 kcal
  Interventions: Drug: Whole Egg
- Healthy Diet (HD) (Active Comparator): 2020-2025 Dietary Guidelines for Americans adherent dietary pattern containing 3 eggs/week/2000 kcal (HD)
  Interventions: Drug: Whole Egg

INTERVENTIONS:
Drug: Whole Egg — Whole Large, Grade A Egg

SUMMARY:
This study will examine the effect of a healthy diet containing 2 eggs per day compared to a healthy diet containing 3 eggs per week on biomarkers of heart health after 4 weeks.

DETAILED DESCRIPTION:
This is a 2-period, randomized, crossover, controlled feeding study examining the effect of 2020-2025 Dietary Guidelines for Americans adherent dietary patterns containing 2 eggs/day/2000 kcal (HD+E) compared to 3 eggs/week/2000 kcal (HD) on biomarkers of cardiovascular health and function after 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* LDL-C ≥115 mg/dL and ≤190 mg/L
* BMI of 25-35 kg/m2
* Intake of <14 eggs/week for the prior 3 months
* Blood pressure <140/90 mmHg
* Fasting blood glucose <126 mg/dL
* Fasting triglycerides <350 mg/dL
* ≤10% change in body weight in the prior 6 months

Exclusion Criteria:

* Type 1 or type 2 diabetes or fasting blood glucose ≥126 mg/dL
* Prescription of anti-hypertensive, lipid lowering or glucose lowering drugs
* Intake of supplements that affect the outcomes of interest and unwilling to cease during the study period
* Diagnosed liver, kidney, or autoimmune disease
* Prior cardiovascular event (e.g., stroke, heart attack)
* Current pregnancy or intention of pregnancy within the next 6 months
* Lactation within prior 6 months
* Follows a vegetarian or vegan diet
* Food allergies/intolerance/sensitives/dislikes of foods included in the study menu
* Antibiotic use within the prior 1 month
* Oral steroid use within the prior 1 month
* Use of tobacco or nicotine containing products with in the past 6 months
* Cancer any site within the past 10 years (eligible if ≥10 years without recurrence) or non-melanoma skin cancer with in the past 5 years (eligible if ≥5 years without recurrence)
* Participation in another clinical trial within 30 days of baseline
* Currently following a restricted or weight loss diet
* Prior bariatric surgery
* Intake of >14 alcoholic drinks/week and/or lack of willingness to consume a maximum of two standard drinks per week while enrolled in the study and/or not willing to avoid alcohol consumption for 48 hour prior to test visits

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 65 (Estimated)
Dates: Start 2024-04-25 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
LDL-cholesterol change | 4 weeks
  Assessed from fasting blood draw expressed in mg/dL. LDL-cholesterol will be measured directly via enzymatic assay. Change in LDL-cholesterol will be calculated as the mean of the end of diet measures (i.e., mean of day 1 and day 2 values) minus the mean of the baseline measures (i.e., mean of day 1 and day 2 values).

SECONDARY OUTCOMES:
Triglyceride change | 4 weeks
  Assessed from fasting blood draw expressed in mg/dL.
Total cholesterol change | 4 weeks
  Assessed from fasting blood draw expressed in mg/dL.
HDL-cholesterol change | 4 weeks
  Assessed from fasting blood draw expressed in mg/dL.
LDL-cholesterol to HDL-cholesterol ratio change | 4 weeks
  LDL-cholesterol and HDL-cholesterol will be measured from a fasting blood draw expressed in mg/dL. The ratio will be calculated as LDL-C divided by HDL-C
Change in particle size and number of LDL, HDL, VLDL and chylomicrons | 4 weeks
  Measured via Nuclear Magnetic Resonance
Change in central systolic and diastolic blood pressure | 4 weeks
  Blood pressure measured assessed using a SphymoCor Xcel (Atcor Medical)
Change in brachial systolic and diastolic blood pressure | 4 weeks
  Blood pressure measured assessed using a SphymoCor Xcel (Atcor Medical)
Change in fasting serum insulin | 4 weeks
  Serum insulin levels assessed in a fasting blood draw and expressed in micro IU/ml
Change in fasting plasma glucose concentration | 4 weeks
  Glucose assessed in a fasting blood draw and expressed in mg/dL
Change in Fructosamine | 4 weeks
  Fructosamine assess in a fasting blood draw and expressed in micro IU/ml
Change in Homeostatic Model Assessment for Insulin Resistance (HOMA-IR) | 4 weeks
  Calculated from insulin and glucose measured from a fasting blood sample. Calculated as (insulin × glucose) / 22.5
Change in carotid-femoral pulse wave velocity | 4 weeks
  A measure of arterial stiffness assessed using a SphymoCor Xcel (Atcor Medical). Expressed in meters/second.
Change in trimethylamine N-oxide (TMAO) | 4 weeks
  Measured in fasting blood. Expressed as µmol/L
Change in choline | 4 weeks
  Measured in fasting blood. Expressed as µmol/L
Change in carnitine | 4 weeks
  Measured in fasting blood. Expressed as µmol/L

OTHER OUTCOMES:
Change in the composition of the gut microbiota | 4 weeks
  Abundance measured using 16 s rRNA sequencing

CONTACTS AND LOCATIONS:
Overall Officials: Kristina Petersen, Principal Investigator — The Pennsylvania State University
Locations (1):
- The Pennylvania State University, University Park, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data will be deposited into an open access repository once results from all pre-specified primary and secondary outcomes are published.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: After publication of all pre-specified primary and secondary outcomes

DOCUMENTS (1):
  • Statistical Analysis Plan (2024-04-11): https://cdn.clinicaltrials.gov/large-docs/00/NCT06120400/SAP_000.pdf